CLINICAL TRIAL: NCT07005661
Title: Multicenter, Prospective, Randomized Controlled Trial of Autologous Platelet Rich Plasma (PRP) Use in Open Surgery for Type A Aortic Dissection
Brief Title: Use of PRP in Open Surgery for Type A Aortic Dissection
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); Xiangya Hospital of Central South University (Other); Guangzhou First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KS2025076; 2023ZD0504400 (Other Grant/Funding Number: the Ministry of Science and Technology of China)
Record Dates: First submitted 2025-05-23; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Aortic Dissection Type A; Transfusions; Platelet Rich Plasma (PRP); Organ Protection
Keywords: aortic dissection; transfusions; platelet rich plasma
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PRP Group (Experimental): Participants in this group will undergo standard blood management and will receive autologous platelet rich plasma (PRP) infusion during open surgery for Type A aortic dissection.
  Interventions: Biological: Autologous Platelet Rich Plasma; Procedure: Standard Blood Management
- Control Group (Active Comparator): Participants in this group will not receive autologous PRP infusion during open surgery for Type A aortic dissection and will undergo standard blood management.
  Interventions: Procedure: Standard Blood Management

INTERVENTIONS:
Biological: Autologous Platelet Rich Plasma — Platelet apheresis was initiated immediately after central venous catheterization and completed before systemic heparinization using the XTRA system (LivaNova, UK). Whole blood was collected at ~60 mL/min via central venous access, ~300 mL per cycle, anticoagulated with sodium citrate. After separation, autologous platelet rich plasma and concentrated RBCs were obtained. The process was repeated for 4-6 cycles, collecting plasma equal to ~20-30% of estimated blood volume (Nadler formula). Crystalloids or colloids were infused during the procedure, and RBCs from the prior cycle were reinfused to maintain hemodynamic stability. Platelet rich plasma was stored in collection bags, agitated at room temperature, and reinfused after heparin neutralization .
  Arms: PRP Group
Procedure: Standard Blood Management — Perioperative transfusion is based on intraoperative hemodynamics and internal environment. Routine blood salvage is performed, with tranexamic acid given throughout (30 mg/kg IV loading dose, 16 mg/kg/h IV maintenance, 2 mg/kg for CPB priming). CPB is primed with 1500 ml using an integrated oxygenator, without ultrafiltration emphasis. At surgery's end, heparin-protamine neutralization is guided by a decision-making system, with point-of-care coagulation monitoring to selectively transfuse blood products based on coagulation abnormalities.

SUMMARY:
The goal of this clinical trial is to determine if autologous platelet rich plasma (PRP) can reduce the need for blood transfusions in patients undergoing open surgery for Type A aortic dissection. It will also evaluate the potential organ-protective effects of autologous PRP. The main questions it aims to answer are:

1. Does PRP reduce the amount of allogeneic red blood cell transfusions for participants?
2. Does PRP administration provide protective effects on organs (heart, liver, lungs, kidneys, brain) in participants?

Researchers will compare the administration of autologous PRP with no PRP infusion to assess whether PRP can reduce blood transfusions and provide organ-protective effects in patients undergoing open surgery for Type A aortic dissection.

Participants will:

1. Receive autologous PRP infusion during surgery
2. Undergo multiple checkups and tests before and after surgery
3. Be recorded for allogeneic red blood cell usage within 24 hours perioperatively and all allogeneic blood products usage during the entire hospitalization
4. Be assessed for organ function (heart, liver, lungs, kidneys, brain) and symptom-related outcomes through clinical evaluations

DETAILED DESCRIPTION:
This multicenter, prospective, randomized, double-blind clinical trial aims to evaluate the efficacy of autologous platelet rich plasma (PRP) in improving outcomes for patients undergoing open surgery for Type A aortic dissection. The study primarily focuses on PRP's ability to reduce transfusion while also exploring its potential role in organ protection. Autologous PRP is prepared from the patient's own blood and administered intraoperatively, integrated with standard blood management practices .

The trial employs a two-arm design, with participants randomly assigned to either the PRP group or the control group. The intervention aligns seamlessly with existing surgical protocols, ensuring feasibility across multiple centers. Data collection emphasizes real-time monitoring and standardized procedures to maintain consistency. The double-blind approach, where participants, investigators, and outcome assessors are masked, minimizes bias and enhances the reliability of results.

The rationale for this trial stems from the high morbidity associated with Type A aortic dissection surgery, particularly due to excessive bleeding and organ injury. Preliminary evidence suggests that PRP may enhance hemostasis and tissue repair, offering a novel therapeutic avenue for this high-risk procedure. This study seeks to provide robust evidence on PRP's clinical utility, potentially shaping future surgical management strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing open surgery for type A aortic dissection (TAAD);
2. Body weight between 60-100 kg; hemoglobin (Hb) > 120 g/L; platelet count (PLT) ≥ 120 × 10⁹/L;
3. Able to understand the purpose of the study, voluntarily participate, and sign the informed consent form.

Exclusion Criteria:

1. Requires mechanical ventilation before surgery;
2. Age under 18 or over 70 years;
3. Use of anticoagulant or antiplatelet drugs within 7 days before surgery;
4. Cardiogenic shock, cardiac arrest, severe hypotension (requiring two or more vasopressors), or mechanical circulatory support within 24 hours before surgery;
5. Renal failure requiring dialysis;
6. Severe coagulopathy or active bleeding tendency;
7. Known history of heparin-induced thrombocytopenia (HIT);
8. Severe psychiatric illness or other conditions affecting study reliability;
9. Any condition deemed unsuitable by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Units of Allogeneic RBC Transfusion Within 24 Hours Perioperatively | From anesthesia induction to 24 hours post-surgery
  The total number of allogeneic RBC units transfused from the start of anesthesia induction through 24 hours post-surgery for Type A aortic dissection, to evaluate the effect of autologous PRP on transfusion .

SECONDARY OUTCOMES:
Total Volume of Allogeneic Blood Products Used During Hospitalization | From anesthesia induction to hospital discharge
  The cumulative volume of allogeneic blood products (including red blood cells, plasma, platelets, and cryoprecipitate) used throughout the entire hospitalization period for Type A aortic dissection surgery, to assess the broader impact of autologous PRP on transfusion.
Intraoperative Blood Loss | From the start of anesthesia induction to the end of surgery.
  Estimated intraoperative blood loss, recorded based on anesthesia records and the surgeon's assessment. This outcome is used to evaluate whether autologous PRP contributes to reduced intraoperative bleeding.
Postoperative 24-Hour Chest Drainage Volume | Within the first 24 hours after surgery
  The total chest drainage volume (mL) within 24 hours after surgery, based on actual measured values. This outcome is used to assess postoperative bleeding and evaluate the potential hemostatic effect of PRP.
Postoperative Cardiac Dysfunction | 24 hours before surgery and 24 hours after surgery
  Defined by elevated cardiac troponin T (cTnT), new ischemic changes on ECG, or reduced ejection fraction on transthoracic echocardiography, compared to preoperative values. This outcome aims to evaluate the potential cardioprotective effect of autologous platelet rich plasma (PRP).
Postoperative Pulmonary Dysfunction | 24 hours before surgery and 24 hours after surgery
  Defined as a decreased PaO₂/FiO₂ ratio or elevated neutrophil elastase levels postoperatively, compared to baseline. This outcome aims to assess the potential effect of PRP on pulmonary function preservation.
Postoperative Intestinal Dysfunction | 24 hours before surgery and 24 hours after surgery
  Defined by increased levels of diamine oxidase (DAO) or intestinal fatty acid-binding protein (I-FABP) postoperatively, compared to preoperative baseline. This outcome is intended to explore the potential protective role of PRP on intestinal barrier function.
Postoperative Renal Dysfunction | 24 hours before surgery and 24 hours after surgery
  Defined by increased serum creatinine (Scr), blood urea nitrogen (BUN), neutrophil gelatinase-associated lipocalin (NGAL), or decreased eGFR, relative to preoperative values. This measure aims to evaluate whether PRP use is associated with reduced postoperative renal dysfunction.
Postoperative Hepatic Dysfunction | 24 hours before surgery and 24 hours after surgery.
  Defined by elevated alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin (TBil) levels postoperatively, relative to preoperative baseline. This outcome assesses the potential hepatic protective effect of PRP.
Postoperative Neurological Dysfunction | 24 hours before surgery and 24 hours after surgery.
  Defined by increased neuron-specific enolase (NSE) levels after surgery or the occurrence of new-onset stroke confirmed by clinical evaluation or imaging. This outcome aims to determine whether PRP contributes to neuroprotection in the early postoperative period.
ICU Length of Stay | From postoperative day 0 (the day of surgery) to ICU discharge,up to 30 days.
  Duration of ICU stay, measured in days, from postoperative day 0 (the day of surgery) to ICU discharge, up to 30 days. This outcome evaluates whether autologous PRP affects postoperative ICU recovery. The time frame excludes any preoperative ICU stays due to unrelated conditions.As immediate postoperative ICU transfer is standard for type A aortic dissection, this period accurately reflects surgery-related ICU recovery.
Total Hospital Length of Stay | From postoperative day 0 (the day of surgery) to hospital discharge, up to 60 days.
  Total duration of hospitalization, measured in days, from postoperative day 0 (the day of surgery) to hospital discharge, up to 60 days. This outcome assesses the impact of autologous PRP on overall recovery and resource utilization. Hospital length of stay will be calculated starting from postoperative day 0, which is defined as the date of surgery, to exclude variability introduced by hospitalization prior to the surgical diagnosis or intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng Wang, PhD, Study Director — Department of Anesthesiology, Beijing Anzhen Hospital

IPD SHARING:
Plan to Share IPD: Yes
Shared materials will include the study protocol and statistical analysis plan (SAP). Data will be available starting 6 months after publication of the primary results and will remain accessible for up to 5 years. Access will be granted to researchers with scientifically valid proposals and a signed data use agreement. Requests should be directed to the principal investigator via the sponsor institution.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available starting 6 months after publication of the primary results and will remain accessible for up to 5 years.
Access Criteria: Access will be granted to researchers with scientifically valid proposals and a signed data use agreement. Requests should be directed to the principal investigator via the sponsor institution.